CLINICAL TRIAL: NCT03342469
Title: Food Additives Effects on EEG Profiles in College Students With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University (Other)
Responsible Party: Principal Investigator, Kathleen Holton, Assistant Professor, American University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-2017-151
Record Dates: First submitted 2017-11-09; First posted 2017-11-17 (Actual); Results first posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Food Additives; Artificial Food Coloring; Diet
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: All ADHD participants and a subgroup of control participants will be exposed to all challenge mixtures (artificial food coloring/placebo, placebo/artificial food coloring) with adequate washout periods between exposures.
Who Masked: Participant, Investigator
Masking Description: The investigators and the participants will be masked as to contents of the chocolate cookies provided during the challenge periods. One research assistant will be unblinded and will not have contact with the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ADHD- Artificial food coloring, then placebo (Experimental): Participants first received 225 mg of the six most common artificial food colors (Red 40, Red 3, Yellow 5, Yellow 6, Blue 1, and Blue 2) mixed in chocolate cookies and consumed consecutively over three days (Monday, Tuesday, Wednesday). After a 4-day washout period, they then received placebo of chocolate cookies and consumed them over three days.
  Interventions: Other: Artificial Food Coloring; Other: Placebo
- ADHD - Placebo, then artificial food coloring (Experimental): Participants first received placebo of chocolate cookies and consumed them over three days. After a 4-day washout period, they then received 225 mg of the six most common artificial food colors (Red 40, Red 3, Yellow 5, Yellow 6, Blue 1, and Blue 2) mixed in chocolate cookies and consumed consecutively over three days (Monday, Tuesday, Wednesday).
  Interventions: Other: Artificial Food Coloring; Other: Placebo
- Controls- Artificial food coloring, then placebo (Experimental): Participants first received 225 mg of the six most common artificial food colors (Red 40, Red 3, Yellow 5, Yellow 6, Blue 1, and Blue 2) mixed in chocolate cookies and consumed consecutively over three days (Monday, Tuesday, Wednesday). After a 4-day washout period, they then received placebo of chocolate cookies and consumed them over three days.
  Interventions: Other: Artificial Food Coloring; Other: Placebo
- Controls - Placebo, then artificial food coloring (Experimental): Participants first received placebo of chocolate cookies and consumed them over three days. After a 4-day washout period, they then received 225 mg of the six most common artificial food colors (Red 40, Red 3, Yellow 5, Yellow 6, Blue 1, and Blue 2) mixed in chocolate cookies and consumed consecutively over three days (Monday, Tuesday, Wednesday).
  Interventions: Other: Artificial Food Coloring; Other: Placebo

INTERVENTIONS:
Other: Artificial Food Coloring — 225mg mixed powdered Artificial Food Coloring (AFC)
Other: Placebo — Placebo chocolate cookies

SUMMARY:
The purpose of this study is to examine the effects of food additives on college students with ADHD. This study could potentially answer an important question which still remains unanswered as to whether certain food additives may be able to cause cognitive and electrical activity changes in college students with and without ADHD. In this context, food additives will be artificial food coloring.

DETAILED DESCRIPTION:
Consent will be obtained at the first visit. Baseline data will be collected on the participants, including height, weight, computerized cognitive functioning, and an EEG recording. Participants will also be taught how to keep a detailed food and symptom diary over the following week. One week later, the participant will return to the lab and turn in the food/symptom diary. All ADHD participants and a subgroup of controls (called extended controls or EC) will be trained on how to follow the dietary intervention. Detailed information on the diet will be given, including food additives to avoid, healthy foods which should be eaten, and shopping tips. For the next two weeks, the participant will follow the dietary intervention at home with access to Dr. Holton to answer any questions. The participant will return to the lab after following the diet for two weeks and assessments (cognitive testing, and EEG) will be completed again along information on dietary compliance will be collected. The third meeting will also mark the beginning of the first challenge period. For the challenges, the participant will consume chocolate cookies every Monday, Tuesday, and Wednesday for two weeks. The cookies may or may not contain artificial food coloring depending on the week. Every Wednesday repeat testing will be completed after the cookies are consumed. The participant will be asked not to take ADHD medication on testing days. After two weeks of challenges the study will be completed. The participant will receive information on their performance and on the study results overall.

ELIGIBILITY:
Inclusion Criteria:

* Generally good health
* 18-24 years old
* Currently attending college
* Physician's diagnosis of ADHD (unless control participant)
* Stable medication dose and frequency for 3 months before the study
* Willing to suspend ADHD medication administration on testing day and the day after testing

Exclusion Criteria:

* Presence of comorbid psychiatric condition other than comorbid depression or anxiety
* Autism
* Severe asthma requiring past hospitalization
* Seizure disorder

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Holton, PhD, Principal Investigator — American University
Locations (1):
- American University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with ADHD and neuro-typical controls were recruited from Jan. 2018 until Oct. 2018 at a Mid-Atlantic University.
Pre-assignment Details: Two-week AFC-free diet to standardize intake before randomization to challenge with AFC relative to placebo.
  Washout period of 4 days between challenge with AFC and placebo.
Groups:
- ADHD- Artificial Food Coloring Challenge First, Then Placebo: A high consumer child dose totaling of 225 mg of the six most common artificial food colors (Red 40, Red 3, Yellow 5, Yellow 6, Blue 1, and Blue 2) will be mixed in chocolate cookies and consumed consecutively over three days (Monday, Tuesday, Wednesday). The chocolate will mask the food coloring. The next week they will received placebo cookies for three days.
  Artificial Food Coloring: Artificial Food Coloring (AFC)
- ADHD- Placebo Challenge First, Then Artificial Food Coloring; Control - Placebo First, Then Artificial Food Coloring: The participants will consume chocolate cookies with no food coloring for three days. The next week a high consumer dose totaling of 225 mg of the six most common artificial food colors (Red 40, Red 3, Yellow 5, Yellow 6, Blue 1, and Blue 2) will be mixed in chocolate cookies and consumed consecutively over three days (Monday, Tuesday, Wednesday).
- Control - Artificial Food Coloring First, Then Placebo: A high consumer child dose totaling of 225 mg of the six most common artificial food colors (Red 40, Red 3, Yellow 5, Yellow 6, Blue 1, and Blue 2) will be mixed in chocolate cookies and consumed consecutively over three days (Monday, Tuesday, Wednesday). The chocolate will mask the food coloring. The next week they will received placebo cookies for three days.
Period: Overall Study
Arm/Group | ADHD- Artificial Food Coloring Challenge First, Then Placebo | ADHD- Placebo Challenge First, Then Artificial Food Coloring | Control - Artificial Food Coloring First, Then Placebo | Control - Placebo First, Then Artificial Food Coloring
Started | 9 | 9 | 3 | 8
Completed | 9 | 8 | 3 | 8
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The ADHD group is college students diagnosed with ADHD and the control group is college students not diagnosed with ADHD. All ADHD participants (except for one drop out before randomization) and 11 controls participants moved on the the randomized placebo-controlled crossover challenge portion of the study.
Groups:
- ADHD Group: College students diagnosed with ADHD.
- Control Group: College students not diagnosed with ADHD
- Total: Total of all reporting groups
Arm/Group | ADHD Group | Control Group | Total
Number analyzed (Participants) | 18 | 11 | 29
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 19.0 [17 to 21] | 20.0 [18 to 22] | 20 [18 to 22]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 21
  Male | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 13 | 8 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 18 | 11 | 29
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 22.26 [15.44 to 29.44] | 24.10 [19.17 to 29.03] | 24.10 [15.44 to 29.44]
GPA [Median (Inter-Quartile Range); unit: GPA] | 3.45 [2.78 to 4.12] | 3.60 [3.14 to 4.06] | 3.5 [2.78 to 4.12]
Adult ADHD Self-Report Scale (ASRS) [Mean (Standard Deviation); unit: units on a scale] — Name: Adult ADHD Self-Report Scale-V1.1 Construct: Self-report checklist of adult ADHD symptoms to screen for possibility of ADHD. It is not meant to be diagnostic. According to the documentation, "The questions in the ASRS v1.1 are consistent with DSM-IV criteria and address the manifestations of ADHD symptoms in adults." Total Range: 0-72 points - higher score indicates more and/or higher frequency of adult ADHD symptoms
  units on a scale | 43.44 (11.3) | 24.49 (8.46) | 30.03 (12.52)
Right Handed [Count of Participants; unit: Participants] | 17 | 11 | 28
Year in College [Count of Participants; unit: Participants]
  Freshman | 11 | 2 | 13
  Sophmore | 3 | 5 | 8
  Junior | 3 | 3 | 6
  Senior | 1 | 1 | 2
Head Injury [Count of Participants; unit: Participants] | 7 | 11 | 18
Concussion [Count of Participants; unit: Participants] | 7 | 7 | 14
Diagnoses [Count of Participants; unit: Participants] — This variable included medical and psychological diagnoses. The most commonly reported diagnoses were anxiety and depression.
  Participants | 6 | 5 | 11
Medication Use [Count of Participants; unit: Participants] | 13 | 8 | 21
Alcohol Use [Count of Participants; unit: Participants] | 18 | 11 | 29
Nicotine Use [Count of Participants; unit: Participants] | 6 | 6 | 12
Marijuana Use [Count of Participants; unit: Participants] | 11 | 6 | 17
Other Substance Use [Count of Participants; unit: Participants] | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Power (EEG) During AFC and Placebo Challenge in ADHD and Control Groups
Description: Electroencephalography (EEG) is an objective measure of brainwave activity that non-invasively records the electrocortical activity emitted from neuronal postsynaptic outputs using small electrodes placed on the head. Quantitative EEG uses techniques to transform electrocortical voltage amplitudes into frequency bands to reflect mental processes in periodicities instead of raw values. These frequency bands can then be compared before/after treatment and/or between groups to better understand how treatment impacts the brain. Resting-state EEG was collected with eyes-closed, but awake, for four minutes
  Frequency bands assessed: delta 1-4Hz, theta 4-7Hz, alpha 8-13Hz, beta 13-30Hz, gamma 30-50Hz Each frequency band was assessed using: mean power (microvolts^2 of a frequency band divided by the length of the frequency band) a
Time Frame: Collected after three days exposure to AFC (on third day) and after three day exposure to placebo (on third day)
Population: Models run for ADHD and control groups, separately.
Measure: Mean (Standard Deviation); unit: Mean Power (microvolts^2)
Groups:
- ADHD- Artificial Food Coloring; Control - Artificial Food Coloring: 225 mg AFC over three days received either the first or second week.
- ADHD- Placebo: Placebo cookies over three days received either the first for second week.
- Control - Placebo: Placebo cookies over three days received either the first or second week.
Arm/Group | ADHD- Artificial Food Coloring | ADHD- Placebo | Control - Artificial Food Coloring | Control - Placebo
Number analyzed (Participants) | 17 | 17 | 11 | 11
Mean Power (microvolts^2)
  Mean Delta Power | 3.19 (1.93) | 3.09 (3.25) | 3.50 (2.13) | 2.13 (1.07)
  Mean Theta Power | 1.96 (2.40) | 1.60 (1.69) | 1.78 (1.27) | 1.54 (1.27)
  Mean Alpha Power | 3.27 (3.19) | 3.17 (2.75) | 3.05 (2.08) | 3.64 (2.48)
  Mean Beta Power | 0.32 (0.23) | 0.25 (0.13) | 0.31 (0.21) | 0.28 (0.17)
  Mean Gamma Power | 0.10 (0.08) | 0.07 (0.04) | 0.10 (0.06) | 0.09 (0.05)
Statistical Analysis 1: Comparison: ADHD- Artificial Food Coloring vs ADHD- Placebo; Difference in Delta Power in ADHD group with and without exposure to AFC. General linear model assessed the impact of treatment (AFC v. placebo) on each EEG frequency band, taking into account order of materials. Dependent variable = Treatment (EEG power during AFC, EEG power during placebo); independent variable = order (AFC/placebo, placebo/AFC) This is a pilot study, thus a power calculation was not done and it was not power to correct for multiple comparisons; Test type: Other; p > 0.05, repeated measures General Linear Model — Significance level </= 0.05. This was chosen due to the small sample size. The p-value is not adjusted for multiple comparisons as this was a pilot study and a power analysis for sample size was not conducted
Statistical Analysis 2: Comparison: ADHD- Artificial Food Coloring vs ADHD- Placebo; Difference in Theta Power in ADHD group with and without exposure to AFC. General linear model assessed the impact of treatment (AFC v. placebo) on each EEG frequency band, taking into account order of materials. Dependent variable = Treatment (EEG power during AFC, EEG power during placebo); independent variable = order (AFC/placebo, placebo/AFC) This is a pilot study, thus a power calculation was not done and it was not power to correct for multiple comparisons; Test type: Other; p > 0.05, repeated measures General Linear Model — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: ADHD- Artificial Food Coloring vs ADHD- Placebo; Difference in Alpha Power in ADHD group with and without exposure to AFC. General linear model assessed the impact of treatment (AFC v. placebo) on each EEG frequency band, taking into account order of materials. Dependent variable = Treatment (EEG power during AFC, EEG power during placebo); independent variable = order (AFC/placebo, placebo/AFC) This is a pilot study, thus a power calculation was not done and it was not power to correct for multiple comparisons; Test type: Other; p > 0.05, repeated measures General Linear Model — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: ADHD- Artificial Food Coloring vs ADHD- Placebo; Difference in Beta Power in ADHD group with and without exposure to AFC. General linear model assessed the impact of treatment (AFC v. placebo) on each EEG frequency band, taking into account order of materials. Dependent variable = Treatment (EEG power during AFC, EEG power during placebo); independent variable = order (AFC/placebo, placebo/AFC) This is a pilot study, thus a power calculation was not done and it was not power to correct for multiple comparisons; Test type: Other; p = 0.08, repeated measures General Linear Model — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: ADHD- Artificial Food Coloring vs ADHD- Placebo; Difference in Gamma Power in ADHD group with and without exposure to AFC. General linear model assessed the impact of treatment (AFC v. placebo) on each EEG frequency band, taking into account order of materials. Dependent variable = Treatment (EEG power during AFC, EEG power during placebo); independent variable = order (AFC/placebo, placebo/AFC) This is a pilot study, thus a power calculation was not done and it was not power to correct for multiple comparisons; Test type: Other; p = 0.05, repeated measures General Linear Model — [p-value comment as in outcome 1, analysis 1]; F(1,14)= 4.55
Statistical Analysis 6: Comparison: Control - Artificial Food Coloring vs Control - Placebo; Difference in Delta Power in control group with and without exposure to AFC. General linear model assessed the impact of treatment (AFC v. placebo) on each EEG frequency band, taking into account order of materials. Dependent variable = Treatment (EEG power during AFC, EEG power during placebo); independent variable = order (AFC/placebo, placebo/AFC) This is a pilot study, thus a power calculation was not done and it was not power to correct for multiple comparisons; Test type: Other; p > 0.05, repeated measures General Linear Model — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Control - Artificial Food Coloring vs Control - Placebo; Difference in Theta Power in control group with and without exposure to AFC. General linear model assessed the impact of treatment (AFC v. placebo) on each EEG frequency band, taking into account order of materials. Dependent variable = Treatment (EEG power during AFC, EEG power during placebo); independent variable = order (AFC/placebo, placebo/AFC) This is a pilot study, thus a power calculation was not done and it was not power to correct for multiple comparisons; Test type: Other; p > 0.05, repeated measures General Linear Model — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Control - Artificial Food Coloring vs Control - Placebo; Difference in Alpha Power in control group with and without exposure to AFC. General linear model assessed the impact of treatment (AFC v. placebo) on each EEG frequency band, taking into account order of materials. Dependent variable = Treatment (EEG power during AFC, EEG power during placebo); independent variable = order (AFC/placebo, placebo/AFC) This is a pilot study, thus a power calculation was not done and it was not power to correct for multiple comparisons; Test type: Other; p > 0.05, repeated measures General Linear Model — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Control - Artificial Food Coloring vs Control - Placebo; Difference in Beta Power in control group with and without exposure to AFC. General linear model assessed the impact of treatment (AFC v. placebo) on each EEG frequency band, taking into account order of materials. Dependent variable = Treatment (EEG power during AFC, EEG power during placebo); independent variable = order (AFC/placebo, placebo/AFC); Test type: Other; p > 0.05, repeated measures General Linear Model — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Control - Artificial Food Coloring vs Control - Placebo; Difference in Gamma Power in control group with and without exposure to AFC. General linear model assessed the impact of treatment (AFC v. placebo) on each EEG frequency band, taking into account order of materials. Dependent variable = Treatment (EEG power during AFC, EEG power during placebo); independent variable = order (AFC/placebo, placebo/AFC) This is a pilot study, thus a power calculation was not done and it was not power to correct for multiple comparisons; Test type: Other; p > 0.05, repeated measures General Linear Model — [p-value comment as in outcome 1, analysis 1]

2. Primary Outcome: Relative Power (EEG) During AFC and Placebo Challenge in ADHD and Control Groups
Description: Electroencephalography (EEG) is an objective measure of brainwave activity that non-invasively records the electrocortical activity emitted from neuronal postsynaptic outputs using small electrodes placed on the head. Quantitative EEG uses techniques to transform electrocortical voltage amplitudes into frequency bands to reflect mental processes in periodicities instead of raw values. These frequency bands can then be compared before/after treatment and/or between groups to better understand how treatment impacts the brain. Resting-state EEG was collected with eyes-closed, but awake, for four minutes
  Frequency bands assessed: delta 1-4Hz, theta 4-7Hz, alpha 8-13Hz, beta 13-30Hz, gamma 30-50Hz Each frequency band was assessed using: relative power (sum of microvolts^2 of a frequency band divided by total power to get a percent)
Time Frame: Collected after three days exposure to AFC (on third day) and after three day exposure to placebo (on third day)
Population: Models run for ADHD and control groups, separately.
Measure: Mean (Standard Deviation); unit: percentage of total power
Arm/Group | ADHD- Artificial Food Coloring | ADHD- Placebo | Control - Artificial Food Coloring | Control - Placebo
Number analyzed (Participants) | 17 | 17 | 11 | 11
percentage of total power
  Relative Delta Power | 0.26 (0.07) | 0.25 (0.08) | 0.27 (0.07) | 0.23 (0.04)
  Relative Theta Power | 0.19 (0.06) | 0.18 (0.05) | 0.20 (0.07) | 0.19 (0.09)
  Relative Alpha Power | 0.40 (0.11) | 0.42 (0.11) | 0.39 (0.10) | 0.44 (0.10)
  Relative Beta Power | 0.16 (0.05) | 0.16 (0.05) | 0.15 (0.04) | 0.15 (0.05)
  Relative Gamma Power | 0.06 (0.03) | 0.05 (0.02) | 0.06 (0.03) | 0.06 (0.03)
Statistical Analysis 1: Comparison: ADHD- Artificial Food Coloring vs ADHD- Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; p > 0.05, repeated measures General Linear Model — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: ADHD- Artificial Food Coloring vs ADHD- Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Other; p > 0.05, repeated measures General Linear Model — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: ADHD- Artificial Food Coloring vs ADHD- Placebo; [analysis description as in outcome 1, analysis 3]; Test type: Other; p = 0.04, repeated measures General Linear Model — [p-value comment as in outcome 1, analysis 1]; F(1.14)= 4.88, p=0.04
Statistical Analysis 4: Comparison: ADHD- Artificial Food Coloring vs ADHD- Placebo; [analysis description as in outcome 1, analysis 4]; Test type: Other; p > 0.05, repeated measures General Linear Model — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: ADHD- Artificial Food Coloring vs ADHD- Placebo; [analysis description as in outcome 1, analysis 5]; Test type: Other; p > 0.05, repeated measures General Linear Model — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Control - Artificial Food Coloring vs Control - Placebo; [analysis description as in outcome 1, analysis 6]; Test type: Other; p > 0.05, repeated measures General Linear Model — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Control - Artificial Food Coloring vs Control - Placebo; [analysis description as in outcome 1, analysis 7]; Test type: Other; p > 0.05, repeated measures General Linear Model
Statistical Analysis 8: Comparison: Control - Artificial Food Coloring vs Control - Placebo; [analysis description as in outcome 1, analysis 8]; Test type: Other; p > 0.05, repeated measures General Linear Model — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Control - Artificial Food Coloring vs Control - Placebo; Difference in Beta Power in control group with and without exposure to AFC. General linear model assessed the impact of treatment (AFC v. placebo) on each EEG frequency band, taking into account order of materials. Dependent variable = Treatment (EEG power during AFC, EEG power during placebo); independent variable = order (AFC/placebo, placebo/AFC) This is a pilot study, thus a power calculation was not done and it was not power to correct for multiple comparisons; Test type: Other; p > 0.05, repeated measures General Linear Model — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Control - Artificial Food Coloring vs Control - Placebo; [analysis description as in outcome 1, analysis 10]; Test type: Other; p > 0.05, repeated measures General Linear Model — [p-value comment as in outcome 1, analysis 1]

3. Primary Outcome: ADHD Symptoms During AFC and Placebo Challenge in ADHD and Control Groups
Description: Name: Adult ADHD Self-Report Scale-V1.1 Construct: Self-report checklist of adult ADHD symptoms to screen for possibility of ADHD. It is not meant to be diagnostic. According to the documentation, "The questions in the ASRS v1.1 are consistent with DSM-IV criteria and address the manifestations of ADHD symptoms in adults." Total Range: 0-72 points - higher score indicates more and/or higher frequency of adult ADHD symptoms
  Sub-scores:
  1. Inattentive: sum of number/frequency of nine questions (taken from full ASRS questionnaire) related to inattention Range: 0-36 - higher score indicates more and/or higher frequency of inattention symptoms
  2. Hyperactive: sum of number/frequency of nine questions (taken from full ASRS questionnaire) related to hyperactivity Range: 0-36 - higher score indicates more and/or higher frequency of hyperactivity symptoms
Time Frame: Collected after three days exposure to AFC (on third day) and after three day exposure to placebo (on third day)
Population: Models run for ADHD and control groups, separately.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- ADHD- Artificial Food Coloring; Control - Artificial Food Coloring: 225 mg of mixed AFC over three days received either the first or second week.
- ADHD - Placebo Challenge; Control - Placebo: Placebo cookies over three days received either the first or second week.
Arm/Group | ADHD- Artificial Food Coloring | ADHD - Placebo Challenge | Control - Artificial Food Coloring | Control - Placebo
Number analyzed (Participants) | 17 | 17 | 11 | 11
score on a scale
  Total ASRS | 42.06 (13.37) | 41.00 (13.03) | 24.63 (9.87) | 23.81 (11.00)
  Inattentive ASRS | 23.76 (7.14) | 22.71 (6.98) | 14.45 (6.06) | 14.27 (8.18)
  Hyperactive ASRS | 18.29 (6.85) | 18.24 (6.49) | 10.18 (4.47) | 9.55 (5.15)
Statistical Analysis 1: Comparison: ADHD- Artificial Food Coloring vs ADHD - Placebo Challenge; Difference in inattentive ASRS in ADHD group with/without exposure to AFC. General linear model assessed the impact of treatment (AFC v. placebo) on each EEG frequency band, taking into account order of materials. Dependent variable = Treatment (inattentive ASRS score during AFC, inattentive ASRS score during placebo); independent variable = order (AFC/placebo, placebo/AFC) This is a pilot study, thus a power calculation was not done and it was not power to correct for multiple comparisons; Test type: Other; p > 0.05, repeated measures General Linear Model — [p-value comment as in outcome 1, analysis 1]; F(1,15) = 3.65, p = 0.08
Statistical Analysis 2: Comparison: ADHD- Artificial Food Coloring vs ADHD - Placebo Challenge; Difference in hyperactive ASRS in ADHD group with/without exposure to AFC. General linear model assessed the impact of treatment (AFC v. placebo) on each EEG frequency band, taking into account order of materials. Dependent variable = Treatment (hyperactive ASRS score during AFC, hyperactive ASRS score during placebo); independent variable = order (AFC/placebo, placebo/AFC) This is a pilot study, thus a power calculation was not done and it was not power to correct for multiple comparisons; Test type: Other; p > 0.05, repeated measures General Linear Model — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: ADHD- Artificial Food Coloring vs ADHD - Placebo Challenge; Difference in total ASRS in ADHD group with/without exposure to AFC. General linear model assessed the impact of treatment (AFC v. placebo) on each EEG frequency band, taking into account order of materials. Dependent variable = Treatment (total ASRS score during AFC, total ASRS score during placebo); independent variable = order (AFC/placebo, placebo/AFC) This is a pilot study, thus a power calculation was not done and it was not power to correct for multiple comparisons; Test type: Other; p > 0.05, repeated measures General Linear Model — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Control - Artificial Food Coloring vs Control - Placebo; inattentive ASRS in control group with/without exposure to AFC. General linear model assessed the impact of treatment (AFC v. placebo) on each EEG frequency band, taking into account order of materials. Dependent variable = Treatment (inattentive ASRS score during AFC, inattentive ASRS score during placebo); independent variable = order (AFC/placebo, placebo/AFC) This is a pilot study, thus a power calculation was not done and it was not power to correct for multiple comparisons; Test type: Other; p > 0.05, repeated measures General Linear Model — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Control - Artificial Food Coloring vs Control - Placebo; Hyperactive ASRS in control group with/without exposure to AFC. General linear model assessed the impact of treatment (AFC v. placebo) on each EEG frequency band, taking into account order of materials. Dependent variable = Treatment (hyperactive ASRS score during AFC, hyperactive ASRS score during placebo); independent variable = order (AFC/placebo, placebo/AFC) This is a pilot study, thus a power calculation was not done and it was not power to correct for multiple comparisons; Test type: Other; p > 0.05, repeated measures General Linear Model — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Control - Artificial Food Coloring vs Control - Placebo; Difference in total ASRS in control group with/without exposure to AFC. General linear model assessed the impact of treatment (AFC v. placebo) on each EEG frequency band, taking into account order of materials. Dependent variable = Treatment (total ASRS score during AFC, total ASRS score during placebo); independent variable = order (AFC/placebo, placebo/AFC) This is a pilot study, thus a power calculation was not done and it was not power to correct for multiple comparisons; Test type: Other; p > 0.05, repeated measures General Linear Model — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: Participants were asked upon each visit how they were feeling and if they had any negative symptoms to report.
Groups:
- Artificial Food Coloring Challenge: ADHD and control participants combined.
  A high consumer child dose totaling of 225 mg of the six most common artificial food colors (Red 40, Red 3, Yellow 5, Yellow 6, Blue 1, and Blue 2) will be mixed in chocolate cookies and consumed consecutively over three days (Monday, Tuesday, Wednesday).
- Placebo Challenge: ADHD and control participants, combined.
  The participants will consume chocolate cookies with no food coloring for three days.
Arm/Group | Artificial Food Coloring Challenge | Placebo Challenge
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29

LIMITATIONS AND CAVEATS:
This pilot study had a small sample size, and was not powered to correct for multiple comparisons. The control group had imperfect randomization of challenge materials (AFC/placebo=3, placebo/AFC=8). Dietary compliance was only measured once.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-23): https://cdn.clinicaltrials.gov/large-docs/69/NCT03342469/Prot_SAP_000.pdf